CLINICAL TRIAL: NCT03790605
Title: Evaluation of the Host Modulating Effects of 1% Curcumin Chips as an Adjunct to Non Surgical Mechanical Debridement in the Treatment of Periodontitis: A Randomised Controlled Clinical Trial
Brief Title: A Clinical Trial to Study the Effect of a Drug, Curcumin in Patients With Periodontitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KLE Society's Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr. Riya Achamma Daniel, Post graduate student, Principal Investigator, Department of Periodontics, KLE Society's Institute of Dental Sciences, Bangalore, KLE Society's Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: riya1curcumin
Record Dates: First submitted 2018-12-19; First posted 2018-12-31 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Periodontitis
Keywords: periodontitis, 1% curcumin chips, host modulation therapy, anti inflammatory effect, interleukin 1 beta
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: Total subjects = 40 INCLUSION CRITERION
  1. Systemically healthy individuals both males and females of 20-60 years
  2. Presence of a minimum of 20 teeth in the oral cavity
  3. Localised periodontal pockets with probing depths greater than 4mm i.e., Periodontitis in its stages 2 and 3, as described by the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions, and published by the American Academy of Periodontology (AAP) EXCLUSION CRITERION
  1 Known allergy to curcumin and/ or hydroxyl propyl methyl cellulose 2 Systemic diseases and/or Inflammatory conditions, Obesity 3 Former or current tobacco users 4 Chronic consumption of alcohol 5 Use of anti-inflammatory drugs and antibiotics over the past 3 months 6 Periodontal therapy in any form, surgical or non surgical in the past 6 months 7 Pregnant and lactating mothers
Who Masked: Participant, Outcomes Assessor
Masking Description: The study design follows a double blinded design where the participant and the outcome assessor are unaware of the intervention to the subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1% curcumin chip (Experimental): Following routine full mouth scaling and root planing within 48 hours, a single chip of 1% curcumin will be placed locally within a single isolated periodontal pocket(the deepest pocket in a patient will be chosen) using a forceps. The patient will be recalled after two weeks for the placement of another chip(second placement)
  Interventions: Drug: 1 % curcumin chip; Procedure: Scaling and root planing
- Placebo chip (Placebo Comparator): Following routine full mouth scaling and root planing within 48 hours, a single placebo chip will be placed locally within a single isolated periodontal pocket (the deepest pocket in a patient will be chosen) using a forceps. The patient will be recalled after two weeks for the placement of another chip (second placement)
  Interventions: Other: Placebo chip; Procedure: Scaling and root planing

INTERVENTIONS:
Drug: 1 % curcumin chip — CURCUMIN CHIP: 4x5x0.5mm chip of 1% curcumin in biodegradable hydroxy propyl methyl cellulose vehicle
  Arms: 1% curcumin chip
Other: Placebo chip — PLACEBO CHIP: 4x5x0.5mm chip (identical to test chip except for the active therapeutic ingredient) in biodegradable hydroxy propyl methyl cellulose vehicle
  Arms: Placebo chip
Procedure: Scaling and root planing — Routine full mouth scaling and root planing within 48 hours will be performed at baseline prior to local placement of the chips

SUMMARY:
The study will follow a parallel arm, randomised, double blinded, placebo controlled design.

There will be two groups Group 1 = receiving 1% curcumin chips after routine scaling and root planing (n=20) Group 2 = receiving placebo chips after routine scaling and root planing (n=20) Clinical parameters: ( Baseline, 4 weeks, 12 weeks) Probing pocket depth, clinical attachment level, gingival index, plaque index Cytokine parameter ( Baseline, 4 weeks) Interleukin 1 beta in GCF

Statistical analysis Repeated measures of ANOVA Paired t-tests

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy individuals
2. Presence of a minimum of 20 teeth in the oral cavity
3. Localised periodontal pockets with probing depths greater than 4mm i.e., Periodontitis in its stages 2 and 3, as described by the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions, and published by the American Academy of Periodontology (AAP)

Exclusion Criteria:

1. Known allergy to curcumin and/ or hydroxyl propyl methyl cellulose
2. Systemic diseases and/or Inflammatory conditions, Obesity
3. Former or current tobacco users
4. Chronic consumption of alcohol
5. Use of anti-inflammatory drugs and antibiotics over the past 3 months
6. Periodontal therapy in any form, surgical or non surgical in the past 6 months
7. Pregnant and lactating mothers

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Cytokine parameter | Change from Baseline to 4 weeks
  Intragroup comparison within each group (1-curcumin group and 2- placebo group) and intergroup comparison between the two groups of levels of interleukin 1 beta in the gingival crevicular fluid quantified by ELISA in picogram per milliliter

SECONDARY OUTCOMES:
Probing pocket depth | Changes from Baseline to 4 weeks and 12 weeks
  Intragroup within each group (1- curcumin group and 2- placebo group) and intergroup comparison between the two groups
Clinical attachment level | Changes from Baseline to 4 weeks and 12 weeks
  Intragroup within each group (1- curcumin group and 2- placebo group) and intergroup comparison between the two groups
Gingival Bleeding Index by Loe and Silness in 1963 | Changes from Baseline to 4 weeks and 12 weeks
  Intragroup within each group ( 1-curcumin group and 2- placebo group) and intergroup comparison between the two group
Plaque index by Silness and Loe in 1964 | Baseline from. 4 weeks, 12 weeks
  Intragroup within each group ( 1- curcumin group and 2- placebo group) and intergroup comparison between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- K L E society's Dental College, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
For the purpose of confidentiality, as will be promised to the participants while signing the informed consent, all individual records except that of the parameters assessed during the study and the photographs taken will remain unshared to the public or fellow researchers